CLINICAL TRIAL: NCT04420728
Title: Closed-Loop Insulin Delivery Postpartum in Mothers With Type 1 Diabetes and Their Babies' Feeding Practices
Brief Title: Closed-Loop Insulin in Mothers With Type 1 Diabetes and Baby Feeding Practices
Acronym: CLIMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Calgary Health Trust (Other); Medtronic (Industry); Ward of the 21st Century (Other)
Responsible Party: Principal Investigator, Lois Donovan, Clinical Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10027445
Record Dates: First submitted 2020-03-24; First posted 2020-06-09 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus Type 1 Pre-Existing; Pregnancy Related; Feeding Behavior; Infant Development
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early auto-mode enabled (Experimental): Auto mode continuous glucose monitoring enabled 2-10 days post-partum
  Interventions: Combination Product: Early auto-mode
- Delayed auto mode enabled (Active Comparator): Auto mode continuous glucose monitoring enabled 12 weeks post-partum
  Interventions: Combination Product: Delayed auto mode

INTERVENTIONS:
Combination Product: Early auto-mode — Participant will be switched to or continue to use the MiniMed 670G insulin pump in manual mode during pregnancy. After the birth of their child, each participant will be randomized to either early auto-mode enabled MiniMed 670G or delayed auto-mode.
  Arms: Early auto-mode enabled
Combination Product: Delayed auto mode — Participant will be switched to or continue to use the MiniMed 670G insulin pump in manual mode during pregnancy. After the birth of their child, each participant will be randomized to either early auto-mode enabled MiniMed 670G or delayed auto-mode.
  Arms: Delayed auto mode enabled

SUMMARY:
This study will is a parallel two-group randomized controlled trial that will use the MiniMed 670G hybrid closed-loop system's continuous glucose monitor (GCM) insulin pump and computer algorithm to deliver insulin when in "auto mode". This study will be conducted in women with type 1 diabetes after delivery of their neonate to see if "auto-mode" improves blood sugar control, episodes of low blood sugar, burden of diabetes self-care, alters baby's weight and feeding patterns, and partner diabetes distress.

DETAILED DESCRIPTION:
Women work very hard prior during pregnancy to try to control their blood sugars. However, after delivery, women often feel they need a rest from the intense effort they have put into diabetes self-care during pregnancy due to the demands of caring for a newborn, breastfeeding, and sleep deprivation. Attention to blood sugar control after delivery remains important because these new factors a may increase the risk of nighttime low blood sugar and unrecognized low blood sugar. Blood sugar has been shown to influence the sugar levels in breastmilk. How this affects the child has not been well study.

The MiniMed 670G hybrid closed-loop system uses a continuous glucose monitor (GCM) insulin pump and computer algorithm to deliver insulin when in "auto mode". The system uses input about the individual's glucose values obtained from the continuous glucose sensor (CGM) to adjust the amount of insulin that is needed between meals and overnight.

Manual mode of the insulin pump delivers insulin based on preprogrammed insulin delivery settings on the insulin pump regardless of the person's glucose levels.

This is a randomized controlled pilot trial followed by an observational cohort study in postpartum women with type 1 diabetes, of the MiniMed 670G hybrid closed-loop insulin delivery system with early 6 to 10 days postpartum) versus delayed (12 weeks postpartum) auto mode enabled MiniMed 670G hybrid closed-loop insulin delivery system. This study will assess the impact of auto mode enabled hybrid closed-loop on glycemic control, occurrence of maternal hypoglycemia, and burden of diabetes self-care, infant weight and feeding practices. The investigators will also assess the acceptability of the auto mode enabled MiniMed 670G during lactation and postpartum and the feasibility of conducting a larger multicentre trial.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 45, with at least a two year duration of type 1 diabetes, on intensive insulin therapy (at least 3 daily insulin injections or insulin pump) with a Hba1c during pregnancy < 9.9 % at study entry who are confirmed by ultrasound, to have a viable singleton pregnancy between 12 and 32 weeks gestation and are not planning to conceive another pregnancy in the first 24 weeks postpartum.

Exclusion Criteria:

* Non-type 1 diabetes
* Any other physical or psychological disease which, in the opinion of the investigator, is likely to interfere with the normal conduct and interpretation of the study results
* Current treatment with drugs known to interfere with glucose metabolism as judged by the investigator such as high dose systemic corticosteroids, non-selective beta-blockers and MAO inhibitors.
* Known or suspected allergy against insulin.
* Women with advanced nephropathy (eGFR<45), severe autonomic neuropathy, uncontrolled gastroparesis or severe proliferative retinopathy, as judged by the investigator, that is likely to interfere with the normal conduct of the study and interpretation of study results.
* Total daily insulin dose of less than 8 or greater than 250 units/day.
* Severe visual or hearing impairment
* Unable to speak and understand English (or French)
* Planning to conceive another pregnancy within the first six months postpartum

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Effect of Auto vs. Manual Mode of MiniMed 670G on Time in Target Range Assessed via CGM | 12 weeks postpartum
  In postpartum women, with type 1 diabetes does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode result in more time in target range (3.9 to 10 mmol/L) assessed by CGM?

SECONDARY OUTCOMES:
Effect of Auto vs. Manual Mode of MiniMed 670G on Time Spent Below Target Range Assessed via CGM | 12 weeks postpartum
  In postpartum women, with type 1 diabetes does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode result in less time spent below target range assessed by CGM (≥15 minutes with CGM glucose <3.9 mmol/L [level 1], 2.8 mmol/L [level 2] assessed by CGM?
Effect of Auto vs. Manual Mode of MiniMed 670G on Time Spent Above Target Range Assessed via CGM | 12 weeks postpartum
  In postpartum women, with type 1 diabetes does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode result in less time above target range > 10 mmol/L assessed by CGM?
Effect of Auto vs. Manual Mode of MiniMed 670G on Glycemic Variability Assessed via CGM | 12 weeks postpartum
  In postpartum women, with type 1 diabetes does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode result in less glycemic variability assessed by CGM?
Effect of Auto vs. Manual Mode of MiniMed 670G on Diabetes Self-Care Assessed via Diabetes Distress Scale 3 | 12 weeks postpartum
  In postpartum women, with type 1 diabetes does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode impact the burden of diabetes self-care, assessed by the Diabetes Distress Scale 3?
Effect of Auto vs. Manual Mode of MiniMed 670G on Quality of Life Assessed via Diabetes Distress Scale 3 and the Hypoglycemia Fear Survey Questionnaire II | 12 weeks postpartum
  In postpartum women, with type 1 diabetes does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode impact the quality of life, assessed by the Diabetes Distress Scale 3 and the Hypoglycemia Fear Survey Questionnaire II?
Effect of Auto vs. Manual Mode of MiniMed 670G on Sleep Assessed via Pittsburgh Sleep Quality Index | 12 weeks postpartum
  In postpartum women, with type 1 diabetes does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode impact sleep, assessed by the Pittsburgh Sleep Quality Index (PSQI)?
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Assess Acceptability of Auto-mode MiniMed 670G via qualitative interviews. | 24 weeks postpartum
  In postpartum women, with type 1 diabetes is use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode, acceptable to patients, their partners and their care providers, assessed via qualitative interviews.
Assess Feasibility of Auto-mode MiniMed 670G via study recruitment, retention and completion rates. | 24 weeks postpartum
  In postpartum women, with type 1 diabetes is use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode, feasibleto patients, their partners and their care providers, assessed by the recruitment, retention and completion rates for this study?

OTHER OUTCOMES:
Effect of Auto vs. Manual Mode of MiniMed 670G on Infant Feeding Practices Assessed via Child Food and Liquid Intake Questionnaire | 12 weeks postpartum
  In postpartum women, with type 1 diabetes does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode impact infant feeding practices? This will be assessed by the Child Food and Liquid Intake questionnaire.
  There is a 3 point scale for questions about child food and liquid intake. There is a 7 point scale for questions about the frequency of breast milk and other liquids in foods.
Impact of Weaning on Total Daily Insulin Requirement on Women who Discontinue Lactation | 24 weeks postpartum
  Among study women that discontinue lactation during the study period what is the impact of weaning on total daily insulin requirements weekly average in the two weeks prior to commencing weaning compared to the two weeks after weaning completed?
Effect of Auto vs. Manual Mode of MiniMed 670G on Sugar Concentrations in Breast Milk Assessed by Liquid Chromatography | 12 weeks postpartum
  In postpartum women with type 1 diabetes, does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode impact sugars (fructose, glucose and lactose) concentration of breast milk. This will be assessed by liquid chromatography-mass spectrometry on expressed breast milk samples.
Effect of Auto vs. Manual Mode of MiniMed 670G on Breast Milk Consumption Assessed by Difference in Infant Weight | 12 weeks postpartum
  In postpartum women with type 1 diabetes, does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode impact volume of breast milk consumed, assessed by the difference in grams of baby weight before and after feeding as measured on an infant weight scale?
Effect of Auto vs. Manual Mode of MiniMed 670G on Infant Weight, Assessed by Weight Measurements | 12 weeks postpartum.
  1d.) In postpartum women with type 1 diabetes, does use of the MiniMed 670G hybrid closed-loop system, enabled with auto mode compared with the MiniMed 670G in manual mode impact infant weight? This will be assessed by measurements taken at time of study followup visits.
Impact of Weaning on Total Daily Insulin Requirement Assessed by Child Food and Liquid Intake Questionnaire | 24 weeks postpartum
  Among study women that discontinue lactation during the study period what is the impact of weaning on total daily insulin requirements weekly average in the two weeks prior to commencing weaning compared to the two weeks after weaning completed, assessed by the Child Food and Liquid Intake questionnaire?

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donovan LE, Bell RC, Feig DS, Lemieux P, Murphy HR, Sigal RJ, Ho J, Virtanen H, Crawford S, Yamamoto JM. Glycaemic patterns during breastfeeding with postpartum use of closed-loop insulin delivery in women with type 1 diabetes. Diabetologia. 2024 Oct;67(10):2154-2159. doi: 10.1007/s00125-024-06227-z. Epub 2024 Jul 19. PMID 39028360